# Is there an immediate effect on pectoralis minor length after performing a prone scapular retraction exercise using typical sets and repetitions in pain free participants?

4/19/2021

**Informed Consent** 

## **Andrews University Informed Consent Form for Participation in the Research Study Entitled:**

Is There an Immediate Effect on Pectoralis Minor Length After Performing a Prone Scapular Retraction Exercise Using Typical Sets and Repetitions in Pain Free Participants

**Primary Researcher** 

**Research Advisor** 

### Andrews University Department of Physical Therapy

#### INFORMED CONSENT FORM

This research study is part of my dissertation project, in partial fulfillment for my doctorate of science in physical therapy degree, at Andrews University, Berrien Springs, Michigan. Your participation in this study is greatly appreciated. If you have any questions or concerns regarding your research rights now or later, please understand that you can contact the Office of Research and Creative Scholarship (Institutional Review Board or IRB) at Andrews University (269)471-6361 or <a href="mailto:research@andrews.edu">research@andrews.edu</a> or <a href="mailto:irb@andrews.edu">irb@andrews.edu</a>.

**Research Title**: Is There an Immediate Effect on Pectoralis Minor Length After Performing a Prone Scapular Retraction Exercise Using Typical Sets and Repetitions in Pain Free Participants

**Purpose of Study:** The purpose of this study is to determine if performing an exercise where the participant actively pulls there shoulder blades back will change the resting length of a muscle in the front of the chest called the pectoralis minor.

**Duration of participation in study**: You will undergo a brief shoulder examination to confirm your eligibility for this study and lessen the risk of shoulder injury from the exercise performed in this study. If the examination shows no sign of shoulder problems you will have your height measured, and then have your pectoralis minor muscle measured by having the ends of a caliper placed at the front of your shoulder and where the third rib attaches to your breast bone (about 3 inches below the collar bone). After the measurement you will perform an exercise while lying on your stomach. You will then have your pectoralis minor muscle measured again. That will conclude your role in the study. The entire procedure is expected to take less than 10 minutes.

**Benefits:** You will benefit from this study by receiving a brief shoulder examination at no monetary cost. At the end of your participation you will also be given a handout with exercises you can perform at home that are believed to retain shoulder health.

By participating in this study you will help rehab professionals such as physical therapists have a greater understanding of how this exercise affects the shoulder girdle. This information will benefit future individuals with shoulder problems.

**Risks:** This study has been designed to have minimal risk to you, but because all exercise and physical evaluation entails some risk, you could possibly experience pain with the shoulder examination or during the exercise. You could also experience soreness in the upper back a day or two after the exercise, a phenomenon called Delayed Onset Muscle Soreness. Because of these risks it is important that you understand you can withdraw from the study at any time without being denied any benefits of the study.

In light of the COVID-19 pandemic extra precautions will be taken to lessen the risk of infection or spread of COVID-19. These precautions include:

• Both the researcher and the participant will wear a face mask covering the nose and mouth

- Social distancing of 6 feet will be observed whenever possible
- The researcher will wash or sanitize his hands between each participant
- The treatment plinth being used will be sanitized between each participant
- Each participant will use a rolled up towel during this investigation, a new towel will be used for each participant
- The participant will be asked if they are experiencing any COVID-19 symptoms before participating in the study and participants who answer yes will not be able to participate

COVID-19 symptoms include; fever (100.4 degrees or greater), chills, sore throat, headache, cough, muscle or body aches, diarrhea (2x in 24 hours), extreme fatigue, shortness of breath or difficulty breathing, new loss of taste/smell, nausea or vomiting (2x in 24 hours), and congestion or runny nose.

I understand that the researchers, the School of Rehabilitation Sciences at Andrews University, and North Idaho Physical Therapy are not liable for any injury incurred during this study. I understand that I'm participating in this study at my own risk.

**Voluntary Participation:** Participation in this study is completely voluntary, refusal to participate will involve no penalty or loss of benefits to which you are otherwise entitled. You may discontinue participation at any time without penalty or loss of benefits to which you may otherwise be entitled.

**Confidentiality:** I understand that my identity in this study will not be disclosed in any published document. All records will be kept secure by the principal investigator. This consent form, a medical history questionnaire, and an ID number to name translator form will have your name on them. All other records will be kept anonymous by using an identity number. The researcher will keep the records for the duration of the study and all forms containing your name will be shredded upon the conclusion of the study.

Whom to Contact: If you have any questions about your rights as a participant in this research, contact my advisor ...; or the primary researcher ... You can also contact the IRB Office at irb@andrews.edu or at (269) 471-6361.

#### By signing below, I indicate that:

- This study has been explained to me
- I have read this document or it has been read to me
- My questions about this research study have been answered satisfactorily
- I have been told that I may ask the researchers any study related questions in the future or contact them in the event of a research-related injury
- I have been told that I may ask Institutional Review Board (IRB) personnel question about my study rights
- I am entitled to a copy of this form after I have read and signed it
- I voluntarily agree to participate in this study
- By signing the consent form, I am hereby giving permission for my participation in this study. If I have any questions or concerns regarding my rights and welfare during participation in the study I understand I can contact IRB at 269-471-6361 or research@andrews.edu or irb@andrews.edu.

| Participant's signature | Date |
|----------------------------|------|
| Participant's name printed | |
| Researcher Signature | Date |